CLINICAL TRIAL: NCT04051229
Title: The Effect of an Exercise Training Program on Metabolic Flexibility in Older Adults With Prediabetes
Brief Title: Exercise Training and Metabolic Flexibility in Prediabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to financial limitations and time commitments, I am requesting the closure of this research
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00058517; 10000441 (Other Grant/Funding Number: Translational Science Center)
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-06

CONDITIONS: PreDiabetes; Sedentary Lifestyle
Keywords: Metabolic Flexibility; Exercise Induced Metabolic Flexibility
MeSH Terms: conditions — Prediabetic State; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be compared to their individual pre-intervention states. All 20 subjects will be placed in the same group and asked to follow the same exercise protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Training Group (Experimental): All 20 participants will be assigned to this arm. These individuals will participate in 6 weeks of a moderate supervised aerobic exercise training program.
  Interventions: Behavioral: 6-week exercise training program; Behavioral: Standardized isoenergetic high fat diet

INTERVENTIONS:
Behavioral: 6-week exercise training program — Participants will walk at 50% Heart Rate Reserve (HRR) 3 to 5 days per week for 6 weeks at the Department of Health and Exercise Science Clinical Research Center under the supervision of study staff.
Behavioral: Standardized isoenergetic high fat diet — Prior to the submaximal exercise testing visits, all participants will be provided with 3 days of a standardized isoenergetic high fat diet (20% of kcals from carbohydrate, 65% fat; 15% protein) to promote lipid oxidation. The meals will be prepared and provided by the Clinical Research Unit of Wake Forest Baptist Health. Participants will pick up 3 days' worth of food and snacks 4 days prior the testing visit. For the 3 days leading up to the visit, participants will eat the provided foods and complete a compliance assessment.

SUMMARY:
The purpose of the study is to determine if a 6-week exercise training program promotes exercise-induced metabolic flexibility, that is, the ability to switch fuel sources for energy, in older prediabetic adults.

DETAILED DESCRIPTION:
This is an investigator initiated single group intervention trial. All participants will receive a 6-week exercise training program with testing occurring before and following the training program. Participants will be provided with 3 days of a high fat diet prior to each of the three testing sessions at the Clinical Research Unit. All who agree to participate will undergo the same intervention.

The goal of this proposal is to study the impact of a 6-week moderate intensity walking training program on exercise induced lipid metabolic flexibility in older adults with prediabetes. Study Investigators will seek to determine if exercise induced lipid oxidation following a high fat diet is increased in trained individuals relative to their baseline.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years of age
* Sedentary prior to the start of the training program (self-reported: less than 30 minutes of exercise for no more than 1 day a week)
* Prediabetes (measured at first screening: HbA1c = 5.7-6.5%)
* Must be able to pick-up and consume study provided foods
* Willingness to provide informed consent and participate in the intervention
* Must obtain transportation to visits and intervention training sessions
* No contraindications for involvement in a moderate exercise training program or exercise testing procedures by self-report

Exclusion Criteria:

* Self-reported diagnosis of a metabolic or chronic disease such as cardiovascular disease, diabetes, Chronic Obstructive Pulmonary Disease, or movement disorders such as Parkinson's disease, Ataxia, Huntington's Disease
* Current or recent (<12 months) treatment for cancer
* Body Mass Index <18.5 or >/30.0 kg/m2
* Tobacco users
* Febrile or chronic infection within study period
* Aversion to testing procedures
* Hypertension, hyperthyroidism, hypothyroidism
* Unwilling to abstain from ingesting caffeine during study testing periods
* Unwilling to withhold medications that affect metabolic rate during testing periods
* Physically active (>30 minutes per day on more than 1 day per week)
* ECGs that indicate cardiac injury or contraindications to treadmill testing
* Allergic or intolerant to any study-provided foods

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Metabolic Rate-Baseline | Baseline
  Metabolic rate will be measured by gas exchange using indirect calorimeter. For the first (baseline test) and second (follow up test 1) time we monitor gas exchange, participants will exercise for 20 minutes at a workload that elicits 50% of maximal oxygen consumption as determined by Graded Exercise Test #1 done before the exercise training program. The third time (follow up test 2), participants will exercise for 20 minutes at a workload that elicits 50% of oxygen consumption as determined by Graded Exercise Test #2 done after the exercise training program.
Metabolic Rate_6 weeks after exercise training program | 6 weeks exercise training program
  Metabolic rate will be measured by gas exchange using indirect calorimeter. For the first (baseline test) and second (follow up test 1) time we monitor gas exchange, participants will exercise for 20 minutes at a workload that elicits 50% of maximal oxygen consumption as determined by Graded Exercise Test #1 done before the exercise training program. The third time (follow up test 2), participants will exercise for 20 minutes at a workload that elicits 50% of oxygen consumption as determined by Graded Exercise Test #2 done after the exercise training program.
Blood collection_lactate Baseline | Baseline
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of lactate. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_lactate follow up 1 | 6 weeks exercise training program
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of lactate. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_lactate follow up 2 | 3-10 days following Follow-Up Test 1
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of lactate. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_glucose baseline | Baseline
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of glucose. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_glucose follow up 1 | 6 weeks exercise training program
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of glucose. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_glucose follow up 2 | 3-10 days following Follow-Up Test 1
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of glucose. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_nonesterified fatty acids | Baseline
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of nonesterified fatty acids. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_nonesterified fatty acids follow up 1 | 6 weeks exercise training program
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of nonesterified fatty acids. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_nonesterified fatty acids follow up 2 | 3-10 days following Follow-Up Test 1
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of nonesterified fatty acids. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_insulin | Baseline
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of insulin. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_insulin follow up 1 | 6 weeks exercise training program
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of insulin. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.
Blood collection_insulin follow up 2 | 3-10 days following Follow-Up Test 1
  At baseline and follow-up testing visits, 6 blood samples at each visit (times 0, 5, 10, 15, 20, and 50) will be obtained for measures of insulin. Blood draws will happen as gas exchange is being measured. 1 tsp of blood will be taken through a catheter at each time point.

SECONDARY OUTCOMES:
VO2 peak | Baseline (Pre-exercise training)
  The gold standard for assessing cardiovascular fitness is exercise capacity as determined from peak volume of oxygen consumption (VO2peak) and treadmill time during a graded exercise test. A physician supervised, individualized ramp treadmill protocol will be performed on each participant. In this protocol, participants walk at a brisk pace with the speed based on their comfort and fitness. For lower fit individuals, the grade will be increased at a rate of 1%/minute, and for higher fit individuals, the grade will be increased at a rate of 2%/minute. The treadmill test will be performed according to guidelines set by the American College of Sports Medicine (ACSM, 2014), to evaluate the subject's cardiovascular response to exercise.
VO2 peak | 6 weeks (Post exercise training)
  The gold standard for assessing cardiovascular fitness is exercise capacity as determined from peak volume of oxygen consumption (VO2peak) and treadmill time during a graded exercise test. A physician supervised, individualized ramp treadmill protocol will be performed on each participant. In this protocol, participants walk at a brisk pace with the speed based on their comfort and fitness. For lower fit individuals, the grade will be increased at a rate of 1%/minute, and for higher fit individuals, the grade will be increased at a rate of 2%/minute. The treadmill test will be performed according to guidelines set by the American College of Sports Medicine (ACSM, 2014), to evaluate the subject's cardiovascular response to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Miller, PhD, Principal Investigator — Wake Forest Department of Health and Exercise Science
Locations (2):
- United States (2):
  - Department of Health and Exercise Science Clinical Research Center, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center Clinical Research Unit, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04051229/ICF_000.pdf